CLINICAL TRIAL: NCT04838535
Title: The Correlation Between Follicular Fluid Raman Spectrum and Embryo Development in Infertile Patients With Polycystic Ovary Syndrome
Brief Title: Follicular Fluid Raman Shifts and IVF Outcomes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: ShangHai Ji Ai Genetics & IVF Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: JIAI E2019-09
Record Dates: First submitted 2021-04-03; First posted 2021-04-09 (Actual); Last update posted 2021-04-09 (Actual); Status verified 2021-04

CONDITIONS: Polycystic Ovary Syndrome; IVF
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PCOS follicular fluid (Other)
  Interventions: Diagnostic Test: Raman spectrum

INTERVENTIONS:
Diagnostic Test: Raman spectrum — The wavelength of the follicular fluids were scaned by Raman spectrum

SUMMARY:
This study intends to collect about 150 cases of follicular fluid samples from PCOS and non-PCOS infertility patients undergoing in vitro fertilization (IVF) or intracytoplasmic sperm injection (ICSI) cycles (in clinical routines).We tend to detect Raman metabolic profile of the follicular fluid of the PCOS and non-PCOS groups, and find the correlation between the metabolic profile of the follicular fluid of PCOS patients and the oocyte quality, IVF outcome and subsequent embryo development are also under investigation. Metabolomics analysis was applied to look for markers of follicular fluid in PCOS patients, and further exploring data and strategies to improve the embryonic development potential and IVF outcome of PCOS patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients fit the Rotterdam criteria for PCOS
* Patients under IVF cycles

Exclusion Criteria:

* Patients with male factors infertility
* Patients with fallopian tube factors infertility

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2019-06-19 (Actual); Primary Completion 2021-06-19 (Estimated); Study Completion 2021-12-19 (Estimated)

PRIMARY OUTCOMES:
Difference between polycystic ovary syndrome and normal follicular fluids | 24 months
  Raman spectrum was applied and the Raman spectrum characteristic absorption peak can be revealed. PCA analysis was used to measure the degree of differential shifts.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoxi Sun, Prof., Study Chair — Shanghai JiAi Genetics & IVF Institute; Jing Fu, Dr., Principal Investigator — Shanghai JiAi Genetics & IVF Institute
Locations (1):
- Shanghai JiAi Genetics and IVF Institute, Shanghai, Shanghai Municipality, China